CLINICAL TRIAL: NCT05003583
Title: The Influence of Contextual and Constitutional Emotional Processes on Speech Motor Control and Speech Motor Learning in Early Childhood Stuttering
Brief Title: Effects of Emotional Processes on Speech Motor Control in Early Childhood Stuttering.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Syracuse University (Other)
Collaborators: National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: R21DC018103 (NIH); R21DC018103-01A1 (NIH)
Record Dates: First submitted 2021-07-22; First posted 2021-08-12 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Stuttering, Childhood
Keywords: stuttering; preschool; motor control; motor learning; emotional processes; behavioral inhibition
MeSH Terms: conditions — Stuttering

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental Condition (Experimental): Speaking while viewing images with negative and neutral valence
  Interventions: Behavioral: Speaking after viewing pictures with negative and neutral valence

INTERVENTIONS:
Behavioral: Speaking after viewing pictures with negative and neutral valence — Speaking Condition 1: 10 age-appropriate pictures from the International Affective Picture System (IAPS; Lang, Bradley & Cuthbert, 2005) will be shown to participants. These pictures are classified as high arousal, negative valence stimuli. Participants will be asked to repeat a simple phrase between picture presentations.
  Speaking Condition 2: A blank screen will be shown to participants in place of pictures. This condition is classified as low arousal, neutral valence. Participants will be asked to repeat a simple phrase between blank screen picture presentations.

SUMMARY:
This study will compare speech variability between preschool-age children who stutter and typically fluent, age-matched peers. Differences in emotional reactivity, regulation and speech motor control have been implicated in stuttering development in children. This study seeks to understand further how these processes interact. Children will repeat a simple phrase after viewing age-appropriate images of either negative or neutral valence to assess speech motor control.

DETAILED DESCRIPTION:
Stuttering is a developmental disorder that emerges in the preschool years as children are undergoing rapid development of their speech, language, and emotional regulation processes. This study aims to understand how speech motor control and emotional processes interact in young children who do and do not stutter.

In Aim 1, the investigators will be observing how speech motor control and learning are affected by emotional (physiological) arousal. High arousal (e.g., stress) has been shown to disrupt highly skilled performances such as in sports and music performance (Yoshie et al., 2009). Parents of children who stutter often report that that exciting or stressful situations lead to increased stuttering in their children. There is little research, however, on how excitement or stress affects fluency in children.

In Aim 2, the investigators will observe how behavioral inhibition plays a role in speech motor control and motor learning in the context of emotional processes. Behavioral inhibition is one aspect of a child's temperament. Temperament refers to self-regulation as well as emotional, motor, and attentional reactivity that differs among individuals. Children with high behavioral inhibition (BI) are hyper-vigilant and more sensitive to new stimuli and negative emotional states. Therefore, the purpose of Aim 2 is to see if children with high BI are more susceptible to contextual emotional processes, therefore affecting speech motor control and learning.

Outcomes will be measured by calculating the variability in speech motor movements (STI). The two groups, children who stutter and age-matched peers who do not stutter, will be compared to see how speech motor control varies between groups and conditions.

ELIGIBILITY:
Inclusion Criteria:

1. English as the primary language of communication.
2. No history of neurological diseases or diagnosed speech-language disorders apart from stuttering.
3. Parent report or direct observation of oral-facial structural abnormalities (such as cleft lip and/or cleft palate).
4. Free of any medications that may affect neural functions (e.g., medications of seizures).
5. Normal hearing acuity (must pass a hearing screening).
6. Normal vision per parent report.

Exclusion Criteria:

1. Failure to meet the inclusionary criteria listed above
2. Parental report of neurodevelopmental disorders (such as autism spectrum disorders)
3. Parental report of vision problems that are not corrected or corrected with glasses.

Ages: 3 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 68 (Actual)
Dates: Start 2021-05-21 (Actual); Primary Completion 2025-09-30 (Actual); Study Completion 2025-09-30 (Actual)

PRIMARY OUTCOMES:
The spatiotemporal index (STI) of lip aperture during a negative valence condition on Day 1 (pretest). | through study completion, an average of 3 weeks
  The spatiotemporal index (STI), a measure of speech coordination developed by Smith and colleagues (e.g., Smith, Goffman, Zelaznik, Ying & McGillem, 1995). It will be employed to quantify speech motor control ability and speech motor learning effects. The STI reflects the degree to which repeated performance of a task produces movement trajectories that converge on a single pattern. Children produce less stable movement trajectories, as reflected in higher values of the STI (e.g. Smith & Goffman, 1998), while adults produce more stable movement trajectories as reflected in lower STI values. The STI of lip aperture (a relative distance between upper and lower lips) will be calculated.
The spatiotemporal index (STI) of lip aperture during a neutral valence condition on Day 1 (pretest). | through study completion, an average of 3 weeks
  The spatiotemporal index (STI), a measure of speech coordination developed by Smith and colleagues (e.g., Smith, Goffman, Zelaznik, Ying & McGillem, 1995). It will be employed to quantify speech motor control ability and speech motor learning effects. The STI reflects the degree to which repeated performance of a task produces movement trajectories that converge on a single pattern. Children produce less stable movement trajectories, as reflected in higher values of the STI (e.g. Smith & Goffman, 1998), while adults produce more stable movement trajectories as reflected in lower STI values. The STI of lip aperture (a relative distance between upper and lower lips) will be calculated.
The spatiotemporal index (STI) of lip aperture during a negative valence condition on Day 2 (retention). | through study completion, an average of 3 weeks
  The spatiotemporal index (STI), a measure of speech coordination developed by Smith and colleagues (e.g., Smith, Goffman, Zelaznik, Ying & McGillem, 1995). It will be employed to quantify speech motor control ability and speech motor learning effects. The STI reflects the degree to which repeated performance of a task produces movement trajectories that converge on a single pattern. Children produce less stable movement trajectories, as reflected in higher values of the STI (e.g. Smith & Goffman, 1998), while adults produce more stable movement trajectories as reflected in lower STI values. The STI of lip aperture (a relative distance between upper and lower lips) will be calculated.
The spatiotemporal index (STI) of lip aperture during a neutral valence condition on Day 2 (retention). | through study completion, an average of 3 weeks
  The spatiotemporal index (STI), a measure of speech coordination developed by Smith and colleagues (e.g., Smith, Goffman, Zelaznik, Ying & McGillem, 1995). It will be employed to quantify speech motor control ability and speech motor learning effects. The STI reflects the degree to which repeated performance of a task produces movement trajectories that converge on a single pattern. Children produce less stable movement trajectories, as reflected in higher values of the STI (e.g. Smith & Goffman, 1998), while adults produce more stable movement trajectories as reflected in lower STI values. The STI of lip aperture (a relative distance between upper and lower lips) will be calculated.

SECONDARY OUTCOMES:
Skin conductance level (SCL) | through study completion, an average of 3 weeks
  Skin conductance level (SCL) measures the activity of the sympathetic branch of the autonomic nervous system. Higher SCL during experimental conditions as compared to the baseline is associated with higher sympathetic nervous system activity and provides physiologic validation of the emotional reactivity differences between the experimental conditions.
Number of phasic skin conductance responses elicited by picture presentations | through study completion, an average of 3 weeks
  Phasic skin conductance responses (SCR) measures the activity of the sympathetic branch of the autonomic nervous system. It is elicited by specific stimuli (in this study, by the pictures presented in the two experimental conditions).Greater number of SCRs elicited by picture presentations during experimental conditions is associated with higher sympathetic nervous system activity and provides physiologic validation of the emotional reactivity differences between the experimental conditions.
Respiratory sinus arrhythmia (RSA) | through study completion, an average of 3 weeks
  Respiratory sinus arrhythmia (RSA) (rhythmic fluctuations in heart rate associated with the respiratory cycle) measures the activity of the parasympathetic branch of the autonomic nervous system. Decreased RSA during the experimental conditions as compared to the baseline provides physiologic validation of the emotional reactivity differences between the experimental conditions.
Executive function (EF) composite score | through study completion, an average of 3 weeks
  Executive function skills will be assessed through behavioral tasks using the NIH Toolbox Early Childhood Cognition Battery (Gershon et al., 2013; Zelazo et al., 2013). The tasks include the Flanker Inhibitory Control and Attention Test to examine inhibitory control, Picture Sequence Memory Test to examine episodic memory, and Dimensional Change Card Sort Test to examine mental flexibility and attention.

CONTACTS AND LOCATIONS:
Overall Officials: Victoria Tumanova, PhD, Principal Investigator — Syracuse University
Locations (1):
- Syracuse University, Department of Communication Sciences and Disorders, Syracuse, New York, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2021-08-06): https://cdn.clinicaltrials.gov/large-docs/83/NCT05003583/ICF_000.pdf